CLINICAL TRIAL: NCT05111691
Title: Does Dry Needling Mediate Cortical Excitability in Patients With Chronic Low Back Pain?
Brief Title: Dry Needling Effects on Cortical Excitability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Woman's University (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); American Academy of Orthopaedic Manual Physical Therapists (Other)
Responsible Party: Principal Investigator, Sharon Wang-Price, Professor, Texas Woman's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2021-370
Record Dates: First submitted 2021-10-15; First posted 2021-11-08 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: All participants will receive the same dry needling intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dry needling (Experimental): Two needles will be inserted on or near the most tender point of the low back. Two additional needles will be inserted on the opposite side at the level of the most tender point regardless of unilateral or bilateral low back pain (LBP). After piercing the skin, the needle will be directed toward the spinous process in a slight inferior-medial angle (approximately 20-30°). Once the needle is inserted, the treating investigator will use a ultrasound scanner to visualize the needle placement and to confirm that needle has reached the deeper layer of the lumbar multifidus (LM) muscle.
  Once the needle placement is confirmed, it will be pulled slightly in and out within the muscle and redirected in small angles for 10 seconds after insertion. The needles will stay (in situ) in the LM for approximately 10 minutes after the insertion and then will be withdrawn.
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Procedure: Dry needling — Dry needling

SUMMARY:
The investigators plan to use a pre-test post-test research design to investigate whether dry needling (DN) has an effect on cortical excitability in patients with chronic low back pain (CLBP), specifically in patients who have developed central sensitization (CS). Therefore, the primary purpose of this study is to examine the immediate effects of a single session of DN on cortical excitability and neurosensory responses in patients CLBP. There are two specific aims: 1) to examine whether a single session of DN will change cortical excitability corresponding to the lumbar multifidus (LM) muscle, and 2) to examine whether a single session of DN will change neurosensory responses to the stimuli applied to the LM muscles.

The investigators also are interested in exploring whether DN has a differential effect on cortical excitability in patients with CLBP who have developed CS vs. those who have not developed CS. Therefore, the secondary purpose of the study is to compare the immediate effects of a single session of DN on cortical excitability between patients with CLBP who have developed central sensitization (CS) and those who do not have CS. The specific aim is to compare cortical excitability corresponding to the LM in participants with and without CS after a single session of DN.

DETAILED DESCRIPTION:
Research Design:

This study will be pre-test post-test trial, in which all eligible participants will receive a single session of dry needling (DN). All outcome measures will be collected before and immediately after a single session of DN.

Procedure:

Eligible participants will be asked to complete an intake form, asking them about their demographic data, including age, gender, height, weight, occupation, past medical history, and questions related to their low back pain (onset, injury mechanism if any, location, duration, type, and nature). Once the participant's eligibility is confirmed, each participant will complete the Central Sensitization Inventory (CSI) questionnaire to assign each participant either in the CS group or non-CS group using the 40 cutoff score of the CSI.

1. Clinical Assessments:

   Each participant will complete 3 self-reported questionnaires before cortical excitability assessment, including pain intensity determined using the Numeric Pain Rating Scale (NPRS), disability determined using the Modified Oswestry Low Back Pain Disability Questionnaire (modified ODI), and quality of life determined by the Patient-Reported Outcomes Measurement Information System® -short form (PROMIS-29). These questionnaires will be used to describe the characteristics of the participants in this study.
2. Cortical Excitability Assessment:

   Three cortical excitability parameters will be collected: amplitudes of motor evoked potentials (MEPs), intracortical facilitation (ICF) values, and short-interval cortical inhibition (SICI) values. Participants will lie in a prone position for the electromyographic (EMG) setup. EMG activity will be collected from the painful side of the L4-5 area. Following the recommendations of the Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles (SENIAM) project, the electrode for the LM will be placed at the L4-5 level, approximately 2-3 cm from the midline, and will be aligned with a line from the posterior superior iliac spine (PSIS) to the interspace between the L1 and L2 spinous process.

   To obtain MEPs of the LM muscle, the M1 (primary motor cortex) will be stimulated while the participant performs a submaximal voluntary contraction. First, the maximum voluntary isometric contractions (MVIC) of the LM will be determined. During the MVIC testing, each participant will perform the maximum upper extremity and trunk lift with the elbows flexed to approximately 90° and shoulders abducted to approximately 120°, and maintain the lift for 3 seconds while resisting against a load applied at the opposite elbow of the painful side by the testing investigator. Two trials each will be performed and the highest root mean square (RMS) of EMG amplitude will be identified. During the cortical excitability assessment, a target line representing ~ 20% of highest RMS value during MVIC will be placed on the real-time EMG monitor while the participant will be asked to maintain the target LM activation by slightly leaning forward and to maintain lumbar lordosis in a seated position.

   Following the MVIC testing, each participant will be seated on a chair for cortical excitability assessment. A "hot spot" will be determined while the participant maintains a 20% submaximal contraction of the LM (i.e., slightly leaning forward and maintain lumbar lordosis). A hot spot is defined as the site at which the largest MEP amplitude is obtained at the lowest TMS stimulation intensity or output (0-100%). The double-cone coil will be positioned over the M1 area opposite to the participant's most painful side. The intensity of TMS stimulation from one TMS stimulator will begin at 35% of stimulator output and then will be increased gradually to yield a MEP from the LM until a 'hot spot' is observed. Next, the active motor threshold (AMT) will be determined. AMT is defined as the stimulation intensity which yields a peak-to-peak amplitude of MEP larger than 200 μV in 5 out of 10 consecutive trials. Once the AMT is determined, the stimulation intensity will be set at 130% of AMT and 10 stimulations will be delivered to the hot spot. The 10 supra-threshold MEP amplitudes (uV) recorded from the LM will be averaged and the average will be used for statistical analysis.

   For the ICF and SICI testing, two stimuli, one conditioning stimulus and one test stimulus, will be generated from two TMS stimulators connected by a coil (BiStim Module, Magstim Co., UK). In ICF, a subthreshold conditioning (second) TMS at the 90% AMT will be delivered to the hot spot 15 ms after a test (first) TMS at the 100% AMT. In SICI, a subthreshold conditioning TMS at 70% AMT will be delivered 2 ms before a test TMS at a supra-threshold test TMS at 120% AMT. For both ICF and SICI, the amplitude of the conditioned MEP will be expressed relative to the amplitude of the corresponding test MEP. Ten trials will be performed for each of the ICF and SICI tests, and the average of the 10 trials will be used for statistical analysis.
3. Quantitative Sensory Tests (QSTs):

   The two QSTs, pressure pain thresholds (PPTs) and conditioned pain modulation (CPM) tests, will be administered after the cortical excitability assessments both before and after the DN intervention. During the PPT, participants will be given a response button to stop testing on their own, and will be instructed to stop the test as soon as the pressure becomes uncomfortable or painful, and not to allow an uncomfortable or painful sensation to continue. Four trials will be tested on the most tender point around L4-5, but the first trial will be counted as a practice trial. The average of the last three trials will be used for statistical analysis.

   For the CPM test, a thermode will be applied to the most tender point of the low back and then heat temperature will increase at 1°/sec to the point until the participant perceives the heat stimuli painful at 6/10 on the numeric pain rating scale (NPRS). Two thermodes which generate heat stimuli at the temperature that the participant rates 6/10 on the NPRS will be used for the CPM testing, one applied to the most tender point of the low back (test stimulus), and the other on the contralateral side of forearm (conditioning stimulus). The NPRS scores will be collected under the two conditions: test stimuli alone and combined test stimuli and conditioning stimuli. The test stimuli will be applied first for 10 seconds and then the conditioning stimuli for 25 seconds, so that the second application of the testing stimuli (for 10 seconds) would occur after 15 seconds of conditioning stimuli.
4. Dry Needling Intervention:

   Two lengths of sterile, disposable, 0.30 mm x 60 mm solid filament needles (Seirin Corp., Shizuoka, Japan) and 0.30 mm x 100 mm solid filament needles (Shanghai Kangnian Medical Device Co., Ltd., Shanghai, China) will be used in the study. The length of the needle for each participant will be selected based on the size of the participant. Two needles will be inserted on or near the most tender point of the low back. Two additional needles will be inserted on the opposite side at the level of the most tender point regardless of unilateral or bilateral LBP. After piercing the skin, the needle will be directed toward the spinous process in a slight inferior-medial angle (approximately 20-30°). Once the needle is inserted, the treating investigator will use ultrasound (US) scanner to visualize the needle placement and to confirm that needle has reached the deeper layer of the LM. Once the needle placement is confirmed, it will be pulled slightly in and out within the muscle and redirected in small angles for 10 seconds after insertion. The needles will stay (in situ) in the LM for approximately 10 minutes after the insertion and then will be withdrawn.
5. Statistical Analysis:

Descriptive statistics will be calculated for participant characteristics as well as baseline outcome measures (amplitudes of MEPs, ICF values, SICI values, PPTs, and CPM scores) of all participants. Independent t-tests will be used to compare the ratio data of participant characteristics, self-reported questionnaires, and baseline outcome measures between the two groups. Chi-square statistics will be used to analyze categorical data of participant characteristics (e.g., sex, side(s) of pain, testing side).

The statistical analysis used to address the three aims with the alpha level is set at 0.05 for all statistical analyses: 1) three paired-t tests or Wilcoxon signed rank tests for the three cortical excitability variables (amplitudes of MEPs, ICF values, and SICI values), respectively, 2) two paired-t tests or Wilcoxon signed rank tests for the two neurosensory variables (PPT and CPM values), respectively, and 3) three 2 (group) x 2 (time) repeated measure ANOVAs to compare CS and non-CS group for the 3 cortical excitability variables, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years of age
* Have chronic low back pain primarily in the L4-5 area that has persisted at least 3 months and has resulted in pain on at least half the days in the past 6 months

Exclusion Criteria:

* Systemic joint disease (e.g. rheumatoid arthritis, psoriasis arthritis)
* Fracture
* Infection
* Tumor
* Neurological disorders (e.g., radiculopathy, myelopathy, cauda equina syndrome)
* Cancer
* Raynaud's disease
* Pregnancy, previous low back surgery
* Immunocompromised disease (e.g., diabetes mellitus, HIV, AIDS, lupus)
* Bleeding disorders (e.g. hemophilia)
* Use of anti-coagulants (e.g. Coumadin)
* A history of significant head trauma
* An electrical, magnetic, or mechanical implantation (e.g. cardiac pacemakers or intracerebral vascular clip)
* A metal implantation in the head and neck areas,
* A history of seizures or unexplained loss of consciousness
* An immediate family member with epilepsy
* Use of seizure threshold lowering medicine
* Current abuse of alcohol or drugs
* A history of psychiatric illness requiring medication controls
* Inability to maintain the testing and treatment positions (i.e., slightly leaning forward while sitting and prone-lying) for 15 minutes at a time

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Amplitude of motor evoked potential | Before and immediately after the intervention
  Amplitude (uV) of motor evoked potential (MEP) will be obtained from the lumbar multifidus muscle during a submaximal contraction (i.e., 20% maximum voluntary isometric contractions) at a stimulus intensity of 130% of active motor threshold (AMT).
  AMT is defined as the transcranial magnetic stimulation intensity which yields a peak-to-peak amplitude of MEP larger than 200 μV in 5 out of 10 consecutive trials.
Intracortical facilitation | Before and immediately after the intervention
  Intracortical facilitation (%) is a ratio of the amplitude of the conditioned MEP relative to the amplitude of the corresponding test MEP. A subthreshold conditioning (second) TMS at the 90% AMT will be delivered 15 ms after a test (first) TMS at the 100% AMT.
Short-interval intracortical inhibition | Before and immediately after the intervention
  Short-interval intracortical inhibition (%) is a ratio of the amplitude of the conditioned MEP relative to the amplitude of the corresponding test MEP. A subthreshold conditioning (first) TMS at 70% AMT will be delivered 2 ms before a test TMS at a supra-threshold test TMS at 120% AMT.

SECONDARY OUTCOMES:
Pressure pain threshold | Before and immediately after the intervention
  Pressure pain threshold (kPa) is a quantitative sensory test, used to measure deep muscular tissue sensitivity to mechanical pressure stimuli. The test determines the amount of pressure over the lumbar multifidus in which a steadily increasing non-painful pressure stimulus turns into a painful pressure sensation.
Conditioned pain modulation | Before and immediately after the intervention
  Conditioned pain modulation (CPM) is the perceived pain intensity for a test stimulus following application of a conditioning stimulus to a remote area of the body. A numerical pain rating scale (NPRS) (0-10) will be used to determine perceived pain intensity. The CPM score will be calculated by subtracting the NPRS score of the test stimulus in the presence of the conditioning stimulus, from the NPRS score of the test stimulus alone. Therefore, the CPM score will range from 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Wang-Price, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: When the summary data are published. Data obtained through this study may be provided to qualified researchers with academic interest in sickle cell anemia. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Result] da Graca-Tarrago M, Deitos A, Patricia Brietzke A, Torres IL, Cadore Stefani L, Fregni F, Caumo W. Electrical Intramuscular Stimulation in Osteoarthritis Enhances the Inhibitory Systems in Pain Processing at Cortical and Cortical Spinal System. Pain Med. 2016 May 1;17(5):877-891. doi: 10.1111/pme.12930. Epub 2015 Sep 23. PMID 26398594
- [Result] Neblett R, Cohen H, Choi Y, Hartzell MM, Williams M, Mayer TG, Gatchel RJ. The Central Sensitization Inventory (CSI): establishing clinically significant values for identifying central sensitivity syndromes in an outpatient chronic pain sample. J Pain. 2013 May;14(5):438-45. doi: 10.1016/j.jpain.2012.11.012. Epub 2013 Mar 13. PMID 23490634
- [Result] Fritz JM, Irrgang JJ. A comparison of a modified Oswestry Low Back Pain Disability Questionnaire and the Quebec Back Pain Disability Scale. Phys Ther. 2001 Feb;81(2):776-88. doi: 10.1093/ptj/81.2.776. PMID 11175676
- [Result] Deyo RA, Katrina Ramsey, Buckley DI, Michaels L, Kobus A, Eckstrom E, Forro V, Morris C. Performance of a Patient Reported Outcomes Measurement Information System (PROMIS) Short Form in Older Adults with Chronic Musculoskeletal Pain. Pain Med. 2016 Feb;17(2):314-24. doi: 10.1093/pm/pnv046. PMID 26814279
- [Result] Masse-Alarie H, Beaulieu LD, Preuss R, Schneider C. Corticomotor control of lumbar multifidus muscles is impaired in chronic low back pain: concurrent evidence from ultrasound imaging and double-pulse transcranial magnetic stimulation. Exp Brain Res. 2016 Apr;234(4):1033-45. doi: 10.1007/s00221-015-4528-x. Epub 2015 Dec 26. PMID 26708518
- [Result] Tsao H, Danneels LA, Hodges PW. ISSLS prize winner: Smudging the motor brain in young adults with recurrent low back pain. Spine (Phila Pa 1976). 2011 Oct 1;36(21):1721-7. doi: 10.1097/BRS.0b013e31821c4267. PMID 21508892
- [Result] Kiesel KB, Uhl T, Underwood FB, Nitz AJ. Rehabilitative ultrasound measurement of select trunk muscle activation during induced pain. Man Ther. 2008 May;13(2):132-8. doi: 10.1016/j.math.2006.10.003. Epub 2007 Jan 2. PMID 17198763
- [Result] Djordjevic O, Konstantinovic L, Miljkovic N, Bijelic G. Relationship Between Electromyographic Signal Amplitude and Thickness Change of the Trunk Muscles in Patients With and Without Low Back Pain. Clin J Pain. 2015 Oct;31(10):893-902. doi: 10.1097/AJP.0000000000000179. PMID 25380224
- [Result] Sung W, Hicks GE, Ebaugh D, Smith SS, Stackhouse S, Wattananon P, Silfies SP. Individuals With and Without Low Back Pain Use Different Motor Control Strategies to Achieve Spinal Stiffness During the Prone Instability Test. J Orthop Sports Phys Ther. 2019 Dec;49(12):899-907. doi: 10.2519/jospt.2019.8577. Epub 2019 Aug 3. PMID 31378122
- [Result] Chesterton LS, Sim J, Wright CC, Foster NE. Interrater reliability of algometry in measuring pressure pain thresholds in healthy humans, using multiple raters. Clin J Pain. 2007 Nov-Dec;23(9):760-6. doi: 10.1097/AJP.0b013e318154b6ae. PMID 18075402
- [Result] Persson AL, Brogardh C, Sjolund BH. Tender or not tender: test-retest repeatability of pressure pain thresholds in the trapezius and deltoid muscles of healthy women. J Rehabil Med. 2004 Jan;36(1):17-27. doi: 10.1080/16501970310015218. PMID 15074434
- [Result] Geva N, Defrin R. Opposite Effects of Stress on Pain Modulation Depend on the Magnitude of Individual Stress Response. J Pain. 2018 Apr;19(4):360-371. doi: 10.1016/j.jpain.2017.11.011. Epub 2017 Dec 11. PMID 29241836
- [Result] Levy D, Abdian L, Dekel-Steinkeller M, Defrin R. Experimental evidence for weaker endogenous inhibition of trigeminal pain than extra-trigeminal pain in healthy individuals. Cephalalgia. 2018 Jun;38(7):1307-1315. doi: 10.1177/0333102417735851. Epub 2017 Oct 9. PMID 28990805
- [Result] Koppenhaver SL, Walker MJ, Su J, McGowen JM, Umlauf L, Harris KD, Ross MD. Changes in lumbar multifidus muscle function and nociceptive sensitivity in low back pain patient responders versus non-responders after dry needling treatment. Man Ther. 2015 Dec;20(6):769-76. doi: 10.1016/j.math.2015.03.003. Epub 2015 Mar 13. PMID 25801100
- [Result] Wang-Price S, Zafereo J, Couch Z, Brizzolara K, Heins T, Smith L. Short-term effects of two deep dry needling techniques on pressure pain thresholds and electromyographic amplitude of the lumbosacral multifidus in patients with low back pain - a randomized clinical trial. J Man Manip Ther. 2020 Dec;28(5):254-265. doi: 10.1080/10669817.2020.1714165. Epub 2020 Jan 17. PMID 31960773
- [Result] Dunning J, Butts R, Mourad F, Young I, Flannagan S, Perreault T. Dry needling: a literature review with implications for clinical practice guidelines. Phys Ther Rev. 2014 Aug;19(4):252-265. doi: 10.1179/108331913X13844245102034. PMID 25143704
- [Result] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, DeLitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Report of the NIH Task Force on research standards for chronic low back pain. J Pain. 2014 Jun;15(6):569-85. doi: 10.1016/j.jpain.2014.03.005. Epub 2014 Apr 29. PMID 24787228
- [Result] Magerl W, Krumova EK, Baron R, Tolle T, Treede RD, Maier C. Reference data for quantitative sensory testing (QST): refined stratification for age and a novel method for statistical comparison of group data. Pain. 2010 Dec;151(3):598-605. doi: 10.1016/j.pain.2010.07.026. Epub 2010 Oct 20. PMID 20965658